CLINICAL TRIAL: NCT01721356
Title: The Neurobiological Basis and Potential Modification of Emotional Intelligence Through Affective / Behavioral Training
Brief Title: Neurobiological Basis of Emotional Intelligence
Acronym: EQ
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, William Killgore, Associate Professor, Mclean Hospital
Other Study IDs: W81XWH-09-1-0730
Record Dates: First submitted 2012-10-31; First posted 2012-11-05 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Emotional Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy individuals: Healthy individuals ranging in age, race, ethnicity, socioeconomic status, and years of education

SUMMARY:
Emotional Intelligence (EI) is defined as the ability to accurately perceive and identify emotions in oneself and others, understand and use emotions to enhance cognitive processes, and effectively manage one's own emotions as well as those of others. Two major approaches to the construct of emotional intelligence have emerged. These two approaches can be broadly defined as the Trait and Ability Approaches. The Trait Approach, which is typically assessed via self-report measures such as that Bar-On Emotional Quotient Inventory, appears to be strongly related to existing models of personality and coping. The other major approach to EI follows an Ability Model, assuming that EI is similar to but distinct from other types of cognitive intelligence, and involves measurement of a variety of skills and abilities related to emotional processing. An understanding of the neurobiological substrate of emotional intelligence is beginning to emerge. One influential theory that is particularly relevant to the neurobiology of emotional intelligence is the "somatic marker hypothesis," yet there still remains a limited understanding of the neurobiological basis of EI. The proposed investigation will attempt to provide the most comprehensive study to date examining the behavioral, psychological, functional, and brain structural correlates of EI. The proposed study will use neuroimaging techniques to examine the relationship between current measures of EI, behavioral expression of emotionally competent capacities, brain functional responses, and structural cerebral organization.

The specific questions to be addressed and their associated hypotheses are:

1. The two major approaches to EI (i.e., Trait vs. Ability) will show only modest, though significant positive correlations with one another.
2. EI Trait measures will be highly correlated with measures of personality but weakly correlated with specific skills such as facial affect identification, emotional decision-making, and affectively based judgments, whereas EI Ability measures will correlate more highly with specific emotional skill measures.
3. During functional MRI affective challenge tasks, EI scores will be negatively correlated with activity within the Somatic Marker Circuitry suggested by Damasio and colleagues (i.e., ventromedial prefrontal cortex, amygdala, insular cortex), as suggested by the neural efficiency hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 18 and 45
* Right handed
* Primary language must be English

Exclusion Criteria:

* Any history of neurological illness, current DSM-IV Axis I disorder, lifetime history of major depression or psychotic disorder, or head injury with loss of consciousness > 30 minutes
* Complicating medical conditions that may influence the outcome of neuropsychological assessment or functional imaging (e.g., HIV)
* Mixed or left-handedness
* Current score of 15 or greater on Beck Depression Inventory
* Abnormal visual acuity that is not corrected by contact lenses
* Metal within the body, claustrophobia, or other contraindications for neuroimaging
* Less than 9th grade education
* Evidence of impaired reading comprehension
* Excess alcohol use (Males: regular intake of 5+ drinks on one occasion or >2 drinks per day on average for past 2 months; Females: 4+ drinks per day or >1 drink per day on average for past 2 months)
* History of alcoholism or substance use disorder
* Use of illicit drugs
* Best of 4 learning trials of Memory Suppression Task Training below 85%
* Indication of invalid responding, potentially including elevated Omission Rate, Inconsistency Index, or Positive/Negative Impression scales on EQi, or elevated Omission Rate or Scatter score on MSCEIT

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Between 70 and 80 healthy, English speaking, right-handed, adults between the ages of 18 and 45 participated. Attempts were made to include equal numbers of men and women to permit the broadest generalization to the population and to permit direct assessment of gender effects, an issue that has received considerable attention recently regarding the neurobiology of affective processes. Subjects were not excluded on the basis of ethnicity, gender, or sexual orientation. Healthy participants were recruited via local advertisements, including email broadcasts such as the Harvard Hospital and Partners Healthcare systems, internet advertisements, and posting of IRB-approved flyers in various community centers. IRB-approved print advertisements were posted in local newspapers.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2009-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Score on ability measure (MSCEIT) of emotional intelligence | Measure administered on the day of the MRI scan

CONTACTS AND LOCATIONS:
Overall Officials: William D Killgore, PhD, Principal Investigator — Mclean Hospital

REFERENCES:
- [Derived] Bajaj S, Raikes AC, Razi A, Miller MA, Killgore WD. Blue-Light Therapy Strengthens Resting-State Effective Connectivity within Default-Mode Network after Mild TBI. J Cent Nerv Syst Dis. 2021 May 19;13:11795735211015076. doi: 10.1177/11795735211015076. eCollection 2021. PMID 34104033